CLINICAL TRIAL: NCT07359794
Title: The Effect of Binaural Drumbeat Listening With Virtual Reality Goggles During Cystoscopy on Pain, Anxiety and Vital Signs
Brief Title: The Effect of Virtual Reality and Binaural Beats on Pain, Anxiety, and Vital Signs During Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Niran Çoban, Asst.Prof., University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NK
Record Dates: First submitted 2026-01-07; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cystoscopy; Binaural Beats; Virtual Reality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality and binaural beat (Experimental): Before cystoscopy During cystoscopy After cystoscopy
  Interventions: Other: Virtual reality headset and binaural beat listening
- Standard care (No Intervention): Before cystoscopy During cystoscopy After cystoscopy

INTERVENTIONS:
Other: Virtual reality headset and binaural beat listening — Nature video and binaural drumming experience with virtual reality headset
  Arms: Virtual reality and binaural beat

SUMMARY:
This study was conducted as a randomized controlled trial to evaluate the effect of nature videos viewed through virtual reality goggles and binaural beat audio played during cystoscopy on pain, anxiety, and vital signs. The study was conducted between September 2025 and December 2025 with 60 patients who applied to the cystoscopy unit of a public hospital in Istanbul and met the inclusion criteria. Patients in the experimental group (n=30) were shown nature videos using virtual reality goggles and listened to binaural beats through headphones, while patients in the control group (n=30) received no intervention other than routine care. Research data were collected using the Patient Introduction Form, Visual Analog Scale, State Anxiety Scale, and Vital Findings Form.

It was determined that nature videos and binaural beats played through virtual reality goggles during cystoscopy reduced patients' pain and anxiety levels and positively affected their vital signs.

DETAILED DESCRIPTION:
Although cystoscopy is a short procedure performed under local anesthesia, its invasive nature can cause pain, anxiety, and physiological stress responses in patients. This can negatively affect the patient's compliance and overall comfort during the procedure. In recent years, it has been reported that distracting, non-pharmacological, and technology-based applications in surgical and interventional procedures are effective in increasing patient comfort. This study was planned and conducted as a randomized controlled trial to evaluate the effect of nature videos viewed through virtual reality (VR) goggles and binaural beats listened to simultaneously during cystoscopy on patients' pain levels, anxiety levels, and vital signs.The study was conducted between September 2025 and December 2025 at the cystoscopy unit of a public hospital in Istanbul. A total of 60 patients scheduled for cystoscopy and meeting the inclusion criteria were enrolled in the study. Patients were randomly assigned to either the experimental (n=30) or control (n=30) group. Patients in the experimental group were shown nature-themed videos through virtual reality glasses and listened to binaural beats through headphones before and during the cystoscopy procedure. No additional interventions were performed on patients in the control group other than the routine care protocol applied in the clinic. Research data were collected using the Patient Introduction Form, which included patient characteristics; the Visual Analog Scale (VAS) to assess pain levels; the State Anxiety Scale to determine anxiety levels; and the Vital Signs Form, which included systolic-diastolic blood pressure, pulse, and respiratory rate. Measurements were taken before, during, and after the procedure.

The research results show that nature videos and binaural beats played through virtual reality goggles during cystoscopy are an effective intervention in reducing patients' pain and anxiety levels and positively affecting physiological parameters. Due to its non-invasive, low-cost, and easy-to-implement nature, this combination is considered to be a complementary nursing practice that can be integrated into clinical applications to enhance patient comfort during short-term procedures such as cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age or older,

  * Male (Due to the shorter and straighter urethra in women and the procedure causing less discomfort, sampling is only included for male patients.),
  * Planned for diagnostic or therapeutic rigid cystoscopy,
  * Undergoing cystoscopy for the first time,
  * Undergoing a cystoscopy procedure that does not require anesthesia,
  * Without any condition that prevents communication,
  * Without any visual impairment or condition that prevents the use of VR glasses,
  * Without mental disability or cognitive impairment,
  * Individuals who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* • Patients with contraindications for cystoscopy (allergic to lidocaine or other agents used, active urinary tract infection, anatomical problems related to the urethra)

  * Patients who have used analgesic (painkiller) medication within 24 hours prior to cystoscopy
  * Patients who will undergo additional manipulation during cystoscopy (Double J catheter placement or removal, bladder biopsy)
  * Patients who did not comply with the study process and conditions were not included in the study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male (Due to the shorter and straighter urethra in women and the procedure causing less discomfort, sampling is only included for male patients.),
Enrollment: 60 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
The Effect of VR and Binaural Beats on Anxiety | 4 month
  State Anxiety Inventory: In this study, the "State Anxiety Inventory (STAI-I)" will be used before and after the mandala coloring to assess patients' situational anxiety. The inventory evaluates how individuals feel at a particular moment. It includes 20 items, each scored from 1 (Not at all) to 4 (Completely), reflecting the intensity of the emotion experienced. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, and 20 are reverse scored. Total scores range from 20 to 80; higher scores indicate greater anxiety. Additionally, the "Trait Anxiety Inventory (STAI-II)" measures general anxiety independent of specific situations, using a similar 20-item structure with frequency-based responses. The full inventory contains 40 items. High scores on either scale indicate higher anxiety levels.Patients completed the questionnaire before and after cystoscopy.
The Effect of VR and Binaural Beats on Pain | 4 month
  Visual Analog Scale: The Visual Analog Scale is a commonly used unidimensional measure for assessing pain intensity. The VAS is a measurement tool ranging from 0 to 10 cm (0 to 100 mm) in length.
  Since the aim of the study is to determine the effect of the non-pharmacological method used on existing pain, VAS will be used to assess pain before, during, and after cystoscopy
The Effect of VR and Binaural Beats on blood pressure | 4 month
  Patients' blood pressure values will be recorded. The effect of non-pharmacological interventions on patients' blood pressure values will be evaluated. Evaluated before, during, and after the cystoscopy
The Effect of VR and Binaural Beats on pulse | 4 month
  Patients' pulse , values will be recorded. The effect of non-pharmacological interventions on patients' pulse values will be evaluated.Evaluated before, during, and after the cystoscopy
The Effect of VR and Binaural Beats on oxygen saturation | 4 month
  Patients' oxygen saturation , values will be recorded. The effect of non-pharmacological interventions on patients' oxygen saturation values will be evaluated.Evaluated before, during, and after the cystoscopy

CONTACTS AND LOCATIONS:
Overall Officials: NİRAN ÇOBAN, Study Director — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xiong J, Jiang X, Cai B, Zhao L, Zhang Q, Luo J. Binaural beats for perioperative anxiety and pain: A systematic review and meta-analysis. Complement Ther Med. 2025 Dec;95:103299. doi: 10.1016/j.ctim.2025.103299. Epub 2025 Oct 30. PMID 41176178
- [Background] Tani A, Vagheggini G, Moretti F, Del Colombo V, Lehle J, Campana S, Labate A, Tomaiuolo F. Binaural Beats Reduce Postoperative Morphine Consumption in Older adults After Total Knee Replacement Surgery. Altern Ther Health Med. 2021 Mar;27(2):27-30. PMID 32412916
- [Background] Ligree N, Nanda S, Morwal S, Garg K. Effect of binaural beat music and noise cancelling headphones on intraoperative anxiety in patients undergoing spinal anaesthesia - A randomised controlled study. Indian J Anaesth. 2023 Jul;67(7):590-594. doi: 10.4103/ija.ija_740_22. Epub 2023 Jul 14. PMID 37601935
- [Background] Öner, N., Le Compte, A., Durumluk Sürekli Kaygı Envanteri El Kitabı, 2. Baskı, Boğaziçi Üniversitesi Yayınları, No:333, 1985.